CLINICAL TRIAL: NCT06681870
Title: A Phase 1 Study of ASP1893 in Participants With Metastatic or Locally Advanced CLDN6-positive Solid Tumors
Brief Title: A Study of ASP1893 in Adults With Advanced CLDN6-positive Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: A business decision was made to not initiate this study.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1893-CL-0101
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: CLDN6-positive Solid Tumor; Ovarian Cancer; Endometrial Cancer; Non-small Cell Lung Cancer; Testicular Cancer; Metastatic or Locally Advanced Solid Tumor Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Carcinoma, Non-Small-Cell Lung; Testicular Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: ASP1893 (Monotherapy) Dose Escalation (Experimental): Participants will receive sequential dose levels of ASP1893 intravenously every 2 weeks or 3 weeks, for a duration of up to 2 years (26 Cycles).
  Interventions: Drug: ASP1893
- Part 2: ASP1893 (Monotherapy) Dose Expansion (Experimental): Participants with select tumor types who have progressed on standard therapies, are no longer eligible for standard therapies or have refused standard approved therapies will receive 1 of 2 dose regimens of ASP1893 from the Dose Escalation phase.
  Interventions: Drug: ASP1893

INTERVENTIONS:
Drug: ASP1893 — Intravenous infusion

SUMMARY:
Before a treatment can be approved for use, clinical studies need to be done. This study is for people with certain types of cancer that have become worse and are difficult to treat. The types of cancer include testicular, ovarian, non-small cell lung cancer, and cancer of the womb (endometrial cancer). The people's cancer will have either spread to other parts of the body (metastatic) or spread to tissue close by (locally advanced).

The cells from these cancers have a protein called Claudin 6 (CLDN6). These cancer cells are known as CLDN6-positive. ASP1893, the study treatment in this study is thought to bind to CLDN6 and a protein found on certain immune cells. This process "tells" the immune system to attack the tumor.

The main aims of the study are to check the safety of ASP1893 in people with these types of cancer, to check if the people can tolerate ASP1893, and to find a suitable dose of ASP1893.

This study will be in 2 parts. In the first part, different small groups of people with testicular cancer, ovarian cancer, non-small cell lung cancer and endometrial cancer will receive lower to higher doses of ASP1893. This will happen one group after another. People who take part in the second part of this study will receive doses of ASP1893 that worked the best in the first part of the study. Different larger groups of people with ovarian cancer, non-small cell lung cancer, and any of the other types of cancer that responded to ASP1893 in the first part of the study will be able to take part in the second part.

In both parts of the study, ASP1893 will be given to people slowly through a tube into a vein. This is called an infusion. This will happen every 2 or 3 weeks. People will continue to receive ASP1893 for up to 1 year, or until their cancer gets worse or they start to have medical problems. People taking part have the option to continue with ASP1893 for another year if the study doctor decides the study treatment is still working well. People in the study can also choose to stop taking part at any time, without giving a reason. During the study, people will visit their study clinic several times for a health check. This includes standard safety checks and reporting any medical problems. Every 8 or 9 weeks, the study doctors will check if each person's cancer has stayed the same or got worse. This will be done by body scans (CT or MRI scans). People will also have their nervous system checked. This includes checking their mental status, reflexes, balance, and coordination. They will also have an eye exam. A tumor sample will be taken during the study and people will have the option of giving a tumor sample after treatment has finished. If people stop the study treatment, they will have follow-up safety checks for up to 1 year after their last dose of ASP1893.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally advanced (unresectable) or metastatic solid tumor which is confirmed by available pathology records or current biopsy.
* For dose escalation (Part 1), the participant must have 1 of the following malignancies:

  * Epithelial ovarian cancer
  * Endometrial cancer (exclude sarcomas)
  * NSCLC (adenocarcinoma only)
  * Testicular cancer
* For dose expansion (Part 2), the participant must have 1 of the following malignancies:

  * Epithelial ovarian cancer
  * NSCLC (adenocarcinoma only)
  * Tumor type for which anti-tumor activity and/or biomarker response was observed during dose escalation.
* Participant has accessible archival tumor sample that is CLDN6 (claudin-6) positive (≥ 1% tumor membrane staining at any intensity [1+]) determined by central IHC (immunohistochemistry) testing. Participants without available tissue should undergo a mandatory biopsy.
* Participant is required to provide tumor tissue at screening/baseline unless participant has accessible archival tumor tissue that is less than 90 days old. If participant does not have accessible archival tumor tissue that is less than 90 days old and is unable to undergo a biopsy due to safety concerns or not medically feasible, enrollment into the study is at the discretion of the medical monitor. Participant should undergo a tumor biopsy during the treatment period as indicated in the Schedules of Assessments.
* Participant has progressed, is intolerant, has refused or there are no standard approved therapies that impart significant clinical benefit (no limit to the number of prior treatment regimens).
* Participant has at least 1 measurable lesion per RECIST v1.1.
* Participant has an ECOG status of 0 or 1.
* Participant who has received radiotherapy must have completed this therapy (including stereotactic radiosurgery) at least 2 weeks prior to study intervention administration. A 1-week washout is permitted for palliative radiation.
* Participant has adequate organ function prior to start of study intervention. If a participant has received a recent blood transfusion, laboratory tests must be obtained ≥ 2 weeks after any blood transfusion.
* Sex and Contraceptive Requirements
* Female participant is not pregnant and at least 1 of the following conditions apply:

  * Not a WOCBP (woman of child bearing potential)
  * WOCBP who has a negative serum pregnancy test and confirmed not pregnant by medical interview at screening and agrees to follow the contraceptive guidance from the time of informed consent through at least 7 months after final study intervention administration.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 5 half-lives (approximately 10 months) after final study intervention administration.
* Female participant must not donate ova starting at first administration of study intervention and throughout the investigational period and for 7 months after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 4 months after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 4 months after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 4 months after final study intervention administration.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study.

Exclusion Criteria:

* Participant weighs < 40 kg.
* Participant has another malignancy for which treatment is required.
* Participant has ongoing toxicity ≥ Grade 2 per the CTCAE (Common Terminology Criteria for Adverse Events) version 5.0 considered clinically significant and attributable to prior antineoplastic therapies.
* Participant has untreated or active CNS metastases. Participant with previously treated CNS (central nervous system) metastases is eligible, if participant is clinically stable and has no evidence of CNS progression by imaging for at least 4 weeks prior to start of study intervention and is not requiring immunosuppressive doses of systemic steroids (equivalent to > 10 mg per day of prednisone) for longer than 2 weeks.
* Participant has an active autoimmune disease. Participant with type 1 diabetes mellitus, endocrinopathies stably maintained on appropriate replacement therapy or skin disorders (e.g., vitiligo, psoriasis or alopecia) not requiring systemic treatment are allowed.
* Participant with a history of or current ILD (interstitial lung disease).
* Participant has an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, any form of substance abuse or psychiatric illness/social situations that would limit compliance with study visits or requirements or a condition that could invalidate communication.
* Participant has a clinically significant abnormal ECG at screening that imposes a safety risk for participation in the study.
* Participant has symptomatic cardiovascular disease within the preceding 12 months including, but not limited to, the following: significant coronary artery disease (e.g., requiring angioplasty or stenting), acute myocardial infarction or unstable angina pectoris < 3 months prior to screening, uncontrolled hypertension, clinically significant arrhythmia or congestive heart failure (New York Heart Association Grade ≥ 2).
* Participant has active or chronic corneal disorders or active ocular conditions requiring ongoing treatment/monitoring, such as uveitis, uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema and/or monocular vision.
* Participant has received a prior allogeneic bone marrow or solid organ transplant.
* Participant has had a major surgical procedure and has not completely recovered within 28 days prior to the start of study intervention.
* Participant with recent positive antigen test for COVID-19 within 10 days prior to study intervention administration. Note: Participant who is asymptomatic after 10 days from the first positive antigen test may be enrolled.
* Participant requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to ASP1893 administration. A participant who uses a physiologic replacement dose of corticosteroids equivalent to 10 mg per day of prednisone or less is allowed, as is receiving a single dose of systemic corticosteroids, or receiving systemic corticosteroids as premedication for radiologic imaging contrast is eligible.
* Participant was discontinued from prior immunomodulatory therapy due to a Grade ≥ 3 toxicity that was mechanistically related (e.g., immune related) to the agent and life threatening.
* Participant is expected to require another form of antineoplastic therapy while on study intervention.
* Participant has received prior anti-CLDN6 and/or TLR (Toll-like receptor) agonist therapy.
* Participant has received a live vaccine against infectious diseases within 28 days prior to initiation of study intervention.
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant is known to have HIV (human immunodeficiency virus) infection. However, participants with HIV infection with CD4+ T-cell counts ≥ 350 cells/µL and no history of AIDS-defining opportunistic infections within the past 6 months are eligible. Note: No HIV testing is required at screening unless mandated per local requirements.
* Participant has any of the following per screening serology test:

  * HAV (hepatitis A virus) antibodies IgM (immunoglobulin M)
  * Positive HBsAg (hepatitis B surface antigen) or detectable HBV DNA (hepatitis B virus deoxyribonucleic acid). Participant with negative HBsAg, positive anti-HBc (hepatitis B core antibody) and negative anti-HBs (hepatitis B surface antibody) are eligible if HBV DNA is undetectable
  * HCV (hepatitis C virus) antibodies unless HCV RNA (ribonucleic acid) is undetectable
* Participant has any condition which makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to ASP1893 or any components of the formulation used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) | Up to 28 days
  A DLT is defined as any event that cannot clearly be attributed to a cause other than ASP1893.
Number of Participants with Adverse Events (AEs) | Up to 26 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Note: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of study intervention. This includes events related to the (study) procedures.
Number of Participants with Serious Adverse Events (SAEs) | Up to 26 months
  An SAE is any untoward medical occurrence in a patient or clinical study participant, that at any dose either results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent or significant disability/incapacity.
Number of Participants with Neurological exam abnormalities | Up to 25 months
  Number of participants with clinically significant neurological exam values.
Number of Participants with Eye Exam Abnormalities | Up to 25 months
  Number of participants with clinically significant eye exam values.
Number of Participants with Laboratory Value abnormalities and/or AEs | Up to 26 months
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with Vital Signs abnormalities and/or AEs | Up to 26 months
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 26 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants with Physical Examination (PE) abnormalities and/or AEs | Up to 25 months
  Number of participants with potentially clinically significant PE values.
Number of Participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status scores | Up to 25 months
  The ECOG scale will be used to assess performance status. Scores range from 0 (fully active) to 5 (dead). Negative change scores represent an improvement. Positive scores represent a decline in performance.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ASP1893 in serum: area under the concentration-time curve from the time of dosing to 14 days after dosing (AUC14d) | Up to 24 months
  AUC14d will be recorded from the PK serum samples collected.
Pharmacokinetics (PK) of ASP1893 in serum: Maximum concentration: Cmax | Up to 24 months
  Cmax of ASP1893 will be recorded from the PK serum samples collected.
Pharmacokinetics (PK) of ASP1893 in serum: Concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 24 months
  Ctrough will be recorded from the PK serum samples collected.
Objective Response Rate (ORR) of ASP1893 per immune-based Response Evaluation Criteria in Solid Tumors (iRECIST) | Up to 36 months
  ORR is defined as the proportion of participants whose best overall response is a confirmed Complete Response (CR) or Partial Response (PR).
Objective Response Rate (ORR) of ASP1893 per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 36 months
  ORR is defined as the proportion of participants whose best overall response is a confirmed Complete Response (CR) or Partial Response (PR).
Duration of Response (DOR) of ASP1893 per iRECIST | Up to 36 months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) or death due to any cause, whichever occurs first.
Duration of Response (DOR) of ASP1893 per RECIST v1.1 | Up to 36 months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented progressive disease (PD) or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) of ASP1893 per iRECIST | Up to 36 months
  DCR is defined as the proportion of participants whose best overall response is rated as confirmed CR, PR or stable disease.
Disease Control Rate (DCR) of ASP1893 per RECIST v1.1 | Up to 36 months
  DCR is defined as the proportion of participants whose best overall response is rated as confirmed CR, PR or stable disease.
Number of Participants with Positive Anti-Drug Antibodies to ASP1893 | Up to 36 months
Changes in Levels of tumor-infiltrating CD4/CD8 lymphocytes | Up to 25 months
  Proportion of participants with changes in infiltration of CD4/CD8 cells

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.